CLINICAL TRIAL: NCT06982599
Title: Effects of Postbiotics on Mood Disorders in Korean Adults: Eight Week, Randomized Double-Blind, Placebo-Controlled, Parallel-Group Clinical Trial
Brief Title: Effects of Postbiotics on Mood Disorders in Korean Adults
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanyang University (Other)
Collaborators: DSM-Firmenich AG (Unknown)
Responsible Party: Principal Investigator, Yongsoon Park, Professor, Hanyang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: POST-LB-KR; HYUIRB-202503-008 (Other: Hanyang University Institutional Review Board)
Record Dates: First submitted 2025-05-01; First posted 2025-05-21 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-09

CONDITIONS: Mood Disorder
Keywords: mood disorder; postbiotics
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- postbiotics (Experimental): 3 capsules/day postbiotics (20 × 10^9 CFU/day) for 8 weeks
  Interventions: Dietary Supplement: postbiotics
- Placebo (Placebo Comparator): 3 capsules/day placebo for 8 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: postbiotics — 3 capsules/day postbiotics (20 × 10^9 CFU/day) for 8 weeks
  Arms: postbiotics
Dietary Supplement: placebo — 3 capsules/day placebo for 8 weeks
  Arms: Placebo

SUMMARY:
This study was conducted to investigate effects of postbiotics on mood disorders in korean adults

DETAILED DESCRIPTION:
This study is an 8-week, randomized, double-blind, placebo-controlled, parallel-group clinical trial. 52 participants were randomly assigned to either the postbiotics intervention group or a placebo group. The study aimed to evaluate the effects of postbiotics on mood disorders in Korean adults, comparing pre- and post-intervention mood profiles.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 19 and 39 years at the time of screening.
* BMI between 18.5 and 30 at the time of screening.
* CES-D (Center for Epidemiologic Studies Depression Scale) score of 16 or higher.
* Ability to access and respond to the survey via an online link.

Exclusion Criteria:

* Participation in any human clinical trial within the past 3 months before screening.
* History of antipsychotic medication treatment within the past 3 months before screening.
* Presence of chronic diseases, including cardiovascular, endocrine, immune, respiratory, hepatobiliary, renal and urological, neurological, musculoskeletal, inflammatory, hematological, oncological, or gastrointestinal disorders.
* Use of medications or health supplements related to gut health and mood disorders (e.g., antibiotics, laxatives, antidiarrheals, prebiotics, probiotics, postbiotics, anxiolytics, antidepressants, etc.) within 1 month prior to participation in the study.
* History of significant hypersensitivity to postbiotics or starch.
* Alcohol addiction, drug abuse, or suspicion of substance misuse.
* Pregnant or breastfeeding women.
* Any other reasons that the study investigator deems the participant unsuitable for participation.

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Estimated)
Dates: Start 2025-10-13 (Actual); Primary Completion 2025-12-21 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Effect of postbiotics on depressive symptoms measured by the Center for Epidemiologic Studies Depression Scale (CES-D), compared with placebo | week 0, week 8
  Epidemiology Research Center Depression Scale (CES-D):
  The Center for Epidemiologic Studies Depression Scale (CES-D) is a widely used 20-item self-reported instrument designed to measure depressive symptom severity in the general population. Each item is rated on a 4-point scale (0 to 3), assessing emotional, somatic, interpersonal, and positive affect domains over the past week. Total scores range from 0 to 60, with higher scores indicating more severe depressive symptoms.
Effect of postbiotics on momentary mood measured by Ecological Momentary Assessment (EMA), compared with placebo | Three consecutive days at baseline (Week 0) and three consecutive days at follow-up (Week 8)
  Ecological Momentary Assessment (EMA) captures real-time mood states by sending brief questionnaires to participants multiple times per day via online links. Each assessment includes six questions related to current mood and mental state, scored on a continuous slider scale from 0 (not at all) to 100 (very much). Higher scores indicate greater severity of negative mood or emotional distress. The average daily score will be calculated and used to assess change from baseline.
Effect of postbiotics on psychological distress measured by the Depression Anxiety Stress Scale-21 (DASS-21), compared with placebo | week 0, week 8
  The Depression Anxiety Stress Scale (DASS-21) is a validated self-report tool containing 21 items, divided equally into three subscales: depression, anxiety, and stress. Each item is rated on a 4-point scale (0 to 3), and subscale scores are summed. Each subscale score ranges from 0 to 21, with higher scores indicating more severe symptoms in the respective domain.

SECONDARY OUTCOMES:
Effect of postbiotics on perceived stress measured by the Perceived Stress Scale (PSS), compared with placebo | Week 0, Week 8
  The Perceived Stress Scale (PSS) is a validated 10-item self-report questionnaire assessing the degree to which situations in one's life are appraised as stressful. Each item is rated on a scale from 0 (never) to 4 (very often), with total scores ranging from 0 to 40. Higher scores indicate greater perceived stress.
Effect of postbiotics on fecal microbiome composition, compared with placebo | Week 0, Week 8
  Fecal samples will be collected for gut microbiota profiling using 16S rRNA gene sequencing. Participants will be asked to provide approximately 0.5 grams of stool in one container, collected within 24 hours prior to the clinic visit. The sample should be stored in a household freezer until delivery, and will be stored at -80°C upon arrival for microbial DNA extraction and analysis.
Effect of postbiotics on fecal metabolites, compared with placebo | Week 0, Week 8
  For metabolite analysis using ultra-performance liquid chromatography-tandem mass spectrometry (UPLC-MS/MS), participants will be asked to provide approximately 0.5 grams of stool in each of two containers. These samples should be collected within 24 hours prior to the clinic visit, frozen at home, and delivered in a frozen state. Upon receipt, samples will be stored at -80°C for metabolomic profiling.
Effect of postbiotics on gastrointestinal symptoms measured by the Irritable Bowel Syndrome Visual Analog Scale (VAS-IBS), compared with placebo | Weekly from Week 0 to Week 8
  The VAS-IBS is a self-report instrument that assesses gastrointestinal symptoms such as abdominal pain, bloating, diarrhea, constipation, and flatulence. Each symptom is rated on a visual analog scale from 0 (very severe) to 100 (very mild). Lower scores indicate more severe symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No